CLINICAL TRIAL: NCT00619749
Title: Polyphenols Rich Fruit Juice Effects on Endothelial Function and Exercise Capacity
Brief Title: Polyphenols and Endothelial Function
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4125
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Sedentary Subjects
MeSH Terms: interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: juice rich in polyphenols
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: juice poor in polyphenols

INTERVENTIONS:
Dietary Supplement: juice rich in polyphenols — juice during 2 weeks
  Arms: 1
Dietary Supplement: juice poor in polyphenols — juice during 2 weeks
  Arms: 2

SUMMARY:
To determine whether fruit juice rich in polyphenols might increase exercise capacity and memory in healthy sedentary subjects.Both parameters might be improved because of the anti-oxidant effects of polyphenols.

ELIGIBILITY:
Inclusion Criteria:

* sedentary

Exclusion Criteria:

* diabetes

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation | 2 years

SECONDARY OUTCOMES:
Exercise, capacity memory | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard geny, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Physiologie et Explorations Fonctionnelles Hôpitaux Universitaires, Strasbourg, France